CLINICAL TRIAL: NCT03150394
Title: A Randomized, Double-blind, Placebo-controlled Study of the Usefulness of the Probiotic 'Lactobacillus Reuteri' in the Therapy of Quadruple Eradication of Helicobacter Pylori Infection in Usual Clinical Practice
Brief Title: Study of the Usefulness of the Probiotic 'Lactobacillus Reuteri' in the Therapy of Quadruple Eradication of Helicobacter Pylori Infection in Usual Clinical Practice.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Luis Fernandez (Other)
Responsible Party: Sponsor-Investigator, Dr. Luis Fernandez, PhD, Hospital Clínico Universitario de Valladolid
Organization: Hospital Clínico Universitario de Valladolid (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VALACT-2017-01
Record Dates: First submitted 2017-05-05; First posted 2017-05-12 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment of quadruple eradication therapy with GASTRUS (Experimental)
  Interventions: Dietary Supplement: GASTRUS
- Treatment of quadruple eradication therapy with PLACEBO (Placebo Comparator)
  Interventions: Other: PLACEBO

INTERVENTIONS:
Dietary Supplement: GASTRUS — Gastrus will be given from the first day of eradication treatment to completion after 30 days of treatment
  Arms: Treatment of quadruple eradication therapy with GASTRUS
Other: PLACEBO — Placebo will be given from the first day of eradication treatment to completion after 30 days of treatment
  Arms: Treatment of quadruple eradication therapy with PLACEBO

SUMMARY:
Helicobacter pylori is a Gram-negative bacterium with a helical bacillus shape that it's able to penetrate and colonize the stomach mucosal lining by infecting it.

The eradication treatment of H. pylori is supported by numerous consensus groups worldwide and it is generally safe and well tolerated. Standard treatment is based on multiple drug regimens. However, its effectiveness has been increasingly compromised due to the emergence of resistant strains, as well as poor adherence to treatment. Therefore, it's proposed a randomized, double-blind, placebo-controlled study whose aims are:

1. Determine whether the combination of two probiotic strains of L reuteri (Gastrus) will improve gastrointestinal symptoms when associated with four-way therapy (of any type).
2. Prove whether supplementation with Gastrus (food supplement) versus Placebo is able to reduce the gastrointestinal adverse effects of quadruple eradication therapy.

They will be determined by the GSRS gastrointestinal symptom scale in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients attended at the clinic visit who present a positive diagnosis of H pylori infection using different diagnostic techniques (C13 breath test, histology, urease and / or H pylori antigen in stools).
* Age between 18 and 65 years

Exclusion Criteria:

* Patients taking other probiotics 4 weeks prior to study start.
* Patients who have previously received eradicating therapy.
* Patients who are treated with NSAIDs, aspirin or other anti-inflammatory drugs either on an occasional basis (one week prior to the study) or on a chronic basis (3 weeks prior to inclusion).
* Patients who have used oral antibiotics two weeks prior to inclusion.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Global score of gastrointestinal symptoms assessed according the GSRS scale | 30 days

SECONDARY OUTCOMES:
Score obtained from each individual gastrointestinal symptom evaluated according the GSRS scale. Percentage of patients completing treatment | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Fernandez Dr. Jesus Barrio, Study Director — Managers study
Locations (2):
- Spain (2):
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital Universitario Río Hortega., Valladolid

IPD SHARING:
Plan to Share IPD: No